CLINICAL TRIAL: NCT05062538
Title: Patient Perspectives in Breast Cancer Care During COVID-19
Brief Title: Cancer Patient Perspectives During COVID-19
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 20-1434.cc
Record Dates: First submitted 2021-09-29; First posted 2021-09-30 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer
Keywords: COVID-19
MeSH Terms: conditions — Breast Neoplasms; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A web-based survey will be emailed to all adult women diagnosed with invasive breast cancer or ductal carcinoma in situ who have been seen as surgical consultations within the last year (06/01/19-06/01/20).

DETAILED DESCRIPTION:
A web-based survey will be emailed to all adult women diagnosed with invasive breast cancer or ductal carcinoma in situ who have been seen as surgical consultations within the last year (06/01/19-06/01/20). This will ensure that patients at various stages of treatment are included, from initial diagnosis into survivorship. This will allow the investigators to assess changes to initial consultations, surgeries, chemotherapy, and radiation, as well as patient perspectives as it relates to these changes.

The web-based surveys will be given via Redcap. The study team will use a validated questionnaire developed at the University of Miami (Penedo, 2020), which includes a combination of multiple-choice questions, Likert scale ratings, and yes/no questions. A list of potential questions is listed below.

A group of patients will be contacted for semi-structured interviews via telephone as well if (1) patients indicate willingness to participate on a separate RedCap survey or (2) if the patient does not respond to this survey. Phone interviews will be recorded and transcribed verbatim. Multiple members of the research team will separately code the information and evaluate for themes.

ELIGIBILITY:
Inclusion Criteria:

* Adult females with diagnosis of invasive breast cancer or ductal carcinoma in situ, seen as surgical consultation between 06/01/19-06/01/20

Exclusion Criteria:

* Males
* Patients with non-cancer diagnoses
* Patients with no history of breast cancer

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Adult females with diagnosis of invasive breast cancer or ductal carcinoma in situ, seen as surgical consultation between 06/01/19-06/01/20
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Number of participants with changes implemented to breast cancer treatment | 12 months
  Number of participants with changes implemented to breast cancer treatment during the COVID-19 pandemic
Number of participants with treatment concerns during COVID-19 pandemic | 12 months
  Patients with treatment concerns during the COVID-19 pandemic
Number of participants with effects of COVID-19 on psychological, social, and physical well-being of breast cancer patients | 12 months
  Number of participants with effects of COVID-19 on psychological, social, and physical well-being of breast cancer patients

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Tevis, Principal Investigator — University of Colorado Health
Locations (1):
- Colorado Research Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No